CLINICAL TRIAL: NCT03394222
Title: Effect of Preoperative Budesonide Inhalation on Arterial Blood Oxygenation and Intrapulmonary Shunt in Patients Received One-lung Ventilation
Brief Title: Effect of Preoperative Budesonide Inhalation on Arterial Blood Oxygenation and Intrapulmonary Shunt During OLV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FujianUnionAnethesia
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: One research assistant was tasked to give the interventional medication in indentical containers to the anesthesiologists(care provider) in charge of the participants for preoperative preparations.Both the participants and care providers were blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Budesonide inhalation group (Experimental): This group of participants were to receive 2mg/4ml of preoperative budesonide inhalation (Khartoum Road NORTH RYDE NSW 2113 Australia. AstraZeneca Pty Ltd) for 10 to 15min.
  Interventions: Drug: preoperative budesonide inhalation
- Normal saline inhalation group (Placebo Comparator): This group of participants were to receive4ml of preoperative normal saline inhalation for 10 to 15min.
  Interventions: Drug: preoperative normal saline inhalation

INTERVENTIONS:
Drug: preoperative budesonide inhalation
  Arms: Budesonide inhalation group
Drug: preoperative normal saline inhalation
  Arms: Normal saline inhalation group

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial to evaluate the effect of preoperative budesonide inhalation on arterial blood oxygenation and intrapulmonary shunt in patients received one-lung ventilation

DETAILED DESCRIPTION:
Population:

The target population comprises all adult aged 45-65 years who was diagnosed lung cancer and to receive video-assist thoracoscopic lobectomy under general anethesia.The study sample will include 50 subjects of both gender and any race or ethnicity.

Procedures:

Eligible and consented patients will be enrolled into the study if all eligibility criteria are met and will be randomly allocated to one of the two study arms:Budesonide inhalation group vs Normal saline inhalation group

Study Duration:

Overall duration of the study is 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45 yr to 65 yr ,height 155-176cm,weight 45-75kg,body mass index(BMI)18-27kg/m2,ASA Physical Status Classifications I to II,left-lateral position during OLV ,normal cardiac and pulmonary function ,and no cardiac,hepatic,renal and endocrine diseases.Diagnosed with uncomplicated lung cancer and was to receive video-assist thoracoscopic lobectomy under general anesthesia.

Exclusion Criteria:

* FEV1/FVC<70%,asthma,chronic obstructive pulmonary disease,acute lung infection,past history of thoracic surgery. preoperative glucocorticoid medication,preoperative chemotherapy,SpO2 kept below 90% for more than 15 minutes during operation,blood transfusion during operation,OLV less than an hour,occurrence of severe complications like allergic shock.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Arterial blood oxygenation | Arterial blood oxygenation was assessed through blood gas analysis before intervention,before OLV ,10 min after OLV,30 min after OLV,60 min after OLV and 10min after two-lung ventilation.
  Arterial blood oxygenation was assessed through blood gas analysis of sample taken from radial artery

SECONDARY OUTCOMES:
Intrapulmonary shunt | Intrapulmonary shunt was assessed through blood gas analysis before intervention,before OLV ,10 min after OLV,30 min after OLV,60 min after OLV and 10min after two-lung ventilation
  Intrapulmonary shunt was assessed through blood gas analysis of sample taken

CONTACTS AND LOCATIONS:
Overall Officials: Wenhua chen, M.D., Principal Investigator — Fujian Medical University Union Hospital